CLINICAL TRIAL: NCT02592122
Title: Airway Responsiveness in Patients With AECOPD Mechanical Ventilation by Inspiratory and Bronchial Dilation Testchronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: snow (Other)
Collaborators: Primary-investigator,Bing Sun (Unknown)
Responsible Party: Sponsor-Investigator, snow, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-10-COPD
Record Dates: First submitted 2015-10-11; First posted 2015-10-30 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Lung Disease,Obstructive
Keywords: Mechanical ventilation; Chronic obstructive pulmonary disease; Airway resistance; Bronchial dilation test
MeSH Terms: conditions — Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atomization inhalation (Active Comparator): First of all, investigators need to give patients to do the test, the result is more than 12% is positive group, less than 12% is negative group.Second, randomly selected into the atomization group
  Interventions: Drug: Salbutamol Aerosol
- Without atomization inhalation (Active Comparator): First of all, investigators need to give patients to do the test, the result is more than 12% is positive group, less than 12% is negative group.Secondly, the random selection is not the atomization group
  Interventions: Drug: No drugs

INTERVENTIONS:
Drug: Salbutamol Aerosol
  Other Names: Ammonium bromide bromide aerosol
  Arms: Atomization inhalation
Drug: No drugs
  Arms: Without atomization inhalation

SUMMARY:
In the patients with COPD mechanical ventilation, the bronchial dilatation is very common. However, the evaluation of the efficacy of the medical examination and other subjective indicators, such as doctors, depends on the doctor's experience; at present, there is no objective evaluation index. For patients with mechanical ventilation, the risk of cross infection can not only increase the risk of cross infection, but also increase the workload of clinical doctors and nurses. Therefore, this study proposes an objective evaluation method to evaluate the response of COPD patients to bronchial dilation. The hypothesis of this study can be used to guide the clinical medication through the test of the bronchus. If the patients with bronchial dilation test positive were used in the test, the patients were not used. In this evaluation method, the changes of airway resistance were measured by the accurate measurement of the patients with inhaled bronchial dilatation.

ELIGIBILITY:
Inclusion Criteria:

* Acute exacerbation of chronic obstructive pulmonary disease
* The mechanical ventilation time of the outdoor endotracheal intubation in the intensive care unit was less than 48 hours

Exclusion Criteria:

* asthma
* has received tracheotomy
* long term mechanical ventilation (which has been accepted for more than 21 days).
* severe pneumonia
* Patients who cannot use a patient with bronchial dilation
* there's a taboo on the use of a sedative.
* refusal to participate in the study
* 48 hours to pull out the tube

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
airway resistance | 1 day
  The first test of bronchial dilatation
Respiratory mechanics index:PEEPi | 1 day

SECONDARY OUTCOMES:
Mechanical ventilation time | 28 days
length of hospital stay | 30 days
Costs of hospitalization expenses | 30 days
Routine blood test:Eosinophilic cells | 7days

CONTACTS AND LOCATIONS:
Overall Officials: Bing Sun, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Department of respiratory and critical care medicine,Beijing Chao-yang Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Li Y, Chen Y, Wang P. Application of impulse oscillometry and bronchial dilation test for analysis in patients with asthma and chronic obstructive pulmonary disease. Int J Clin Exp Med. 2015 Jan 15;8(1):1271-5. eCollection 2015. PMID 25785124